CLINICAL TRIAL: NCT00199173
Title: Comparison Hepatic Intra-arterial Injection of Yttrium-90 Versus 5FU in Colorectal Cancer Metastatic to the Liver Only
Brief Title: Comparing Hepatic Intra-arterial Injection of Yttrium-90 Microspheres Versus Fluorouracil (5FU) in Colorectal Cancer Metastatic to the Liver Only
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Institut Jules Bordet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sir-Spheres1
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Neoplasm; Secondary Malignant Neoplasm of Liver
Keywords: colorectal cancer; liver metastasis; intraarterial hepatic injection; yttrium loaded microspheres; colorectal neoplasm metastatic to the liver
MeSH Terms: conditions — Colorectal Neoplasms

INTERVENTIONS:
Device: SIR Spheres intra-arterial hepatic

SUMMARY:
This is a Phase III trial comparing hepatic intra-arterial injection of Yttrium-90 microspheres (selective internal radiation [SIR] spheres) versus infusional intravenous (IV) 5FU in colorectal cancer metastatic to the liver only and refractory to standard IV chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma, metastatic to the liver only.
* Failure of prior chemotherapy for advanced colorectal cancer.
* Adequate laboratory values of hematologic, renal and liver function
* World Health Organization (WHO) performance status (PS) <= 2
* Written consent

Exclusion Criteria:

* Pregnant or lactating patients
* Other tumor type than adenocarcinoma (leiomyosarcoma; lymphoma).
* Patients with cirrhosis or other chronic liver disease
* Thrombosis of the hepatic main artery of the portal vein
* Lung shunting > 20% as determined by nuclear medicine breakthrough scan
* Patients with serum bilirubin > 1.0 x upper limit of normal (ULN) or with AST and/or ALT and/or alkaline phosphatase > 5 x ULN
* Patients with concurrent or within 4 week period administration of any other experimental drugs.
* Other serious illness or medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hendlisz, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium